CLINICAL TRIAL: NCT06770335
Title: Strategy-based Cognitive Rehabilitation with Integrated Fatigue Management for Patients with Paediatric Brain Tumour (PBT): an Acceptability and Feasibility Study of the Fatigue, Learning and Memory Enrichment (FLaME) Intervention
Brief Title: The FLaME Cognitive Rehabilitation Study for Childhood Brain Tumour
Acronym: FLaME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Success Charity (Unknown); Child Brain Injury Trust (Unknown); Cambridge University Hospitals NHS Foundation Trust (Other); The UCL Great Ormond Street Institute of Child Health (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22BO24
Record Dates: First submitted 2024-12-24; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Childhood Brain Tumor; Childhood Brain Tumors; Pediatric Brain Neoplasms; Pediatric Brain Tumor
Keywords: Paediatric brain tumour; cognitive rehabilitation; cognition; fatigue; feasibility; acceptability; neuropsychology; neurocognitive; childhood brain tumour
MeSH Terms: conditions — Fatigue | interventions — Educational Status; CASP8 and FADD-Like Apoptosis Regulating Protein

STUDY DESIGN:
Intervention Model Description: The feasibility study employs a randomised, parallel arm design with a standard care control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive rehabilitation with fatigue management (Experimental): A 12-week block of intervention (strategy-based cognitive rehabilitation with fatigue management)
  Interventions: Behavioral: THE FATIGUE, LEARNING, AND MEMORY ENRICHMENT (FLaME) INTERVENTION - Full intervention
- Cognitive rehabilitation only (Experimental): A 6-week block of intervention (strategy-based cognitive rehabilitation alone)
  Interventions: Behavioral: THE FATIGUE, LEARNING, AND MEMORY ENRICHMENT (FLaME) INTERVENTION - Cognitive rehabilitation only
- Standard care (No Intervention): Standard care only

INTERVENTIONS:
Behavioral: THE FATIGUE, LEARNING, AND MEMORY ENRICHMENT (FLaME) INTERVENTION - Full intervention — A novel strategy-based cognitive rehabilitation intervention that can be delivered with or without cognitive fatigue management. Skills are targeted sequentially based on a developmental hierarchical model where cognitive fatigue can be addressed first, followed by adult-supported compensatory strategies, with independent use of strategies for specific impairments delivered only once these earlier levels have been addressed. The 'FLaME' program incorporates strategies that have been trialled and found successful in fatigue (e.g., pacing and activity scheduling) and cognitive rehabilitation (e.g., chunking, elaborative encoding techniques) interventions for children. The intervention address two key issues: 1) to deliver strategy-based cognitive rehabilitation as an alternative to prevailing drill-based approaches, and 2) to integrate fatigue management to improve feasibility and acceptability of cognitive rehabilitation. This arm include the full intervention.
  Arms: Cognitive rehabilitation with fatigue management
Behavioral: THE FATIGUE, LEARNING, AND MEMORY ENRICHMENT (FLaME) INTERVENTION - Cognitive rehabilitation only — A novel strategy-based cognitive rehabilitation intervention that can be delivered with or without cognitive fatigue management. Skills are targeted sequentially based on a developmental hierarchical model where cognitive fatigue can be addressed first, followed by adult-supported compensatory strategies, with independent use of strategies for specific impairments delivered only once these earlier levels have been addressed. The 'FLaME' program incorporates strategies that have been trialled and found successful in fatigue (e.g., pacing and activity scheduling) and cognitive rehabilitation (e.g., chunking, elaborative encoding techniques) interventions for children. The intervention address two key issues: 1) to deliver strategy-based cognitive rehabilitation as an alternative to prevailing drill-based approaches, and 2) to integrate fatigue management to improve feasibility and acceptability of cognitive rehabilitation. This arm includes the cognitive rehabilitation only.
  Arms: Cognitive rehabilitation only

SUMMARY:
Medical treatments have improved survival rates for children with brain tumours. However, most children experience long-term difficulties with 'cognition' (thinking skills such as memory and paying attention) and cognitive fatigue (excessive mental tiredness) after treatment. Thinking difficulties and fatigue can affect a child's ability to learn, and their social and emotional wellbeing. National guidance recommends treatment called 'cognitive rehabilitation' which teaches skills to improve or manage cognitive difficulties. Families often request this, but it is not usually available due to little research. Fatigue may also get in the way of children using and benefiting from cognitive rehabilitation. No research study has offered a fatigue treatment for children recovering from brain tumours. The study aims to see if it is practical and helpful to families to provide cognitive rehabilitation for children affected by brain tumours. The treatment focuses on strategies to help cognition. The investigators will see if adding strategies to manage fatigue helps. The study will include thirty-six 7-17-year-olds who have been treated for brain tumour at Great Ormond Street Hospital. All participants will have had an assessment describing cognitive strengths and weaknesses as part of usual care. Participants will be randomly allocated to one of three groups: 1) cognitive rehabilitation with fatigue management (12 weeks), 2) cognitive rehabilitation only (6 weeks), or 3) usual care. Each child and their carer will complete questionnaires before, during, and after the treatment, and an interview at the end of the treatment. This information will help the researchers see if families find the treatment helpful and practical to take part in, and if adding fatigue strategies is beneficial. Researchers will look at information such as the number of appointments attended, feedback about the treatment, and information about fatigue levels, cognition, and wellbeing. The findings will be used to develop a UK-wide study.

DETAILED DESCRIPTION:
Treatment advances for childhood brain tumour in recent decades have substantially improved mortality rates but come at significant cost to the child's cognitive abilities, alongside the effects of the tumour itself. Up to 100% of children treated for a brain tumour experience some degree of cognitive difficulty despite most having achieved typical cognitive development prior to diagnosis. In most cases the child will experience multiple cognitive difficulties (e.g., with memory, attention, and speed of processing) that severely impact quality of life, mental health, access to education, academic and vocational attainment, and progress towards becoming an independent adult. These cognitive difficulties often emerge and become more severe over time (called 'late effects'). These difficulties have been frequently found in research studies and have informed a strong emphasis on the need for neurorehabilitation in national guidance for childhood brain tumour (e.g. NICE, 2005). Interventions aimed to address cognitive difficulties and support children to resume their developmental trajectory as closely as possible are clearly paramount. However, recent evidence finds that the recommendation for neurorehabilitation is rarely implemented, with cognitive rehabilitation almost entirely unavailable. Poor adherence to national guidance is compounded by the very limited research into cognitive rehabilitation interventions for children treated for brain tumour. The few interventions tried have also had poor feasibility of implementation (e.g., low completion rates) and low acceptability for patients and families.

Cognitive rehabilitation interventions typically involve either 1) 'massed drill-based' practice (sometimes called 'brain training') on cognitive training tasks where the individual repeats a cognitive training exercises over many sessions such as remembering an array of dots; 2) strategy-based approaches which teach strategies to optimise cognition (e.g., memory techniques such as mnemonics), and/or 3) external compensatory aids (e.g., visual reminders). There are few studies of cognitive rehabilitation for children with brain tumour, particularly good quality trials. A small number of studies have focused on drill-based rehabilitation, however, the feasibility and acceptability for this approach for children with brain tumour is low and has well documented problems in poor generalisation to skills beyond the repetitively trained task and poor maintenance of improvements. Rehabilitation in childhood brain injury has greatest potential when it includes cognitive strategy-use, is adapted for developmental level, involves systemic support, and empowers children to develop their own strategies. There is currently one good quality trial of a cognitive rehabilitation intervention that incorporates strategy-use for children with brain tumour. The intervention resulted in improvements in academic attainments and parental report of child attention skills, but with small effect sizes. The program also included a demanding drill-based practice component (requiring 50 hours in total), with only 60% of participants completing the intervention. A subsequent study omitted the drill-based practice and extended the strategy-use component, combining it with parent and teacher strategy support in a smaller pilot study. The power and generalisability of the findings are limited by a small sample size, however some improvements for cognition were found. Parents and children also rated high levels of satisfaction, particularly because the intervention improved their understanding of their cognitive strengths and weakness. Despite some promising findings for strategy-based cognitive rehabilitation, poor feasibility continues to be reflected in low completion rates. No cognitive rehabilitation intervention has addressed the high prevalence of cognitive fatigue (extreme mental tiredness) for children with brain tumours that could predictably limit engagement and completion of interventions. Despite strong recommendations a targeted intervention has yet to be developed for cognitive fatigue for children with brain tumours.

The research was designed to answer two key questions where there is a substantial evidence gap: 1) is a novel strategy-based cognitive rehabilitation intervention acceptable and feasible to children treated for brain tumour and their families, and 2) does adding fatigue management to the intervention improve feasibility and acceptability. The intervention is called The Fatigue, Learning and Memory Enrichment [FLaME] programme. The findings will tell us about the feasibility, acceptability, and preliminary outcomes of the FLaME programme. That is, it will tell us if there are any barriers to putting this intervention in place for young people with brain tumours, how acceptable they find it, and what the level of demand and satisfaction there is with the intervention. We will also seek preliminary information about intervention effectiveness to inform the optimum outcome measurement. This information will inform progress to a larger scale randomised controlled trial (RCT) to meet a substantial evidence gap in an under-researched group. There has been no cognitive rehabilitation trial for childhood brain tumour in the UK before, including within the National Health Service.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 7 years to 17 years, 11 months.
2. Received diagnosis and/or treatment/surveillance at GOSH for a childhood tumour that involved the CNS (brain) and/or oncology treatment to brain.
3. Received or receiving a neuropsychological assessment/consultation at GOSH over the course of the study period or in the 48 months prior to the study period, or under active surveillance with the neuro-oncology multidisciplinary team during the study period.
4. At least 6 months post-diagnosis/acute treatment (surgery and/or radiotherapy), and 3 months post-return to school, with stable disease.
5. One or more scores outside of normal limits (i.e. 1 SD above or below the mean in the direction indicating difficulty) in at least one neuropsychological domain (on performance-based tests or questionnaire-based rating scales).
6. Report impairment (z-score > -0.67) in fatigue on one or more subscales of the PedsQL Multidimensional Fatigue Scale.
7. Capacity/competence of patient or parent/carer to provide informed

Exclusion Criteria:

1. Completed or having another targeted formal psychological intervention for cognitive rehabilitation or fatigue in the past 6 months.
2. Sensorimotor (e.g., visual-motor) impairment only on neuropsychological assessment without additional cognitive difficulty.
3. Current substance misuse from self-report.
4. Currently receiving formal psychiatric care for a diagnosed mental health disorder (including active suicidal ideation), excluding ADHD treatment (if a child has a diagnosis of ADHD they should be treated).
5. Intellectual Disability based on a standard score of more than 2 standard deviations below the mean on a general adaptive behaviour composite and, where available, the General Ability Index of intellect.
6. Patient and parent/carer is unable to communicate verbally and in written form in English.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Goal Based Outcome for management of fatigue | From enrolment to week 14
  The GBO tool is a way of evaluating progress towards goals in clinical work with children, young people, and their families and carers. The GBO compares how far a child or young person feels they have moved towards reaching a goal that they have set for themselves at the beginning of an intervention, on a scale between 0 and 10. 1-3 therapeutic goals are developed collaboratively with a psychologist
Goal Based Outcome for management of cognitive difficulty | From enrolment to week 14
  The GBO tool is a way of evaluating progress towards goals in clinical work with children, young people, and their families and carers. The GBO compares how far a child or young person feels they have moved towards reaching a goal that they have set for themselves at the beginning of an intervention, on a scale between 0 and 10. 1-3 therapeutic goals are developed collaboratively with a psychologist

SECONDARY OUTCOMES:
Multidimensional Fatigue Scale | From enrolment to week 14
  A self-report symptom-specific instrument to measure fatigue in patients with acute and chronic health conditions. Multiple dimensions of fatigue are measured including general fatigue, sleep/rest fatigue, and cognitive fatigue.
Individual daily fatigue analogue scale | From enrolment to week 14
  Rating of subjective fatigue from 0-10 (0 = no fatigue, 10 = severe fatigue) for the morning and afternoon
% School attendance | From enrolment to week 14
  UK Govt. method: each day = 2 sessions and averaged per term and conventional threshold of >=10% of sessions missed as persistent absence)
Behaviour Rating Inventory of Executive Function, Second Edition (BRIEF2) | From enrolment to week 14
  The BRIEF2 screens for executive function skills/difficulties in children and adolescents ages 5 to 18 years. Three domains evaluate cognitive, behavioural, and emotional regulation, and a Global Executive Composite score provides and overall evaluation of executive functioning
Paediatric Quality of Life Inventory (PedsQL) Core + Brain Tumour Module Cognitive Problems scale | From enrolment to week 14
  The core PedsQL is a brief measure of health-related quality of life in children and young people and includes scales on physical functioning, emotional functioning, social functioning, and school functioning. Additional modules can be added for common quality of life difficulties in specific health populations. The Brain Tumour module includes a cognitive problems scale of seven items on the specific cognitive difficulties young people with brain tumours frequently report.
The Brief Illness Perceptions Questionnaire (BIPQ) | From enrolment to week 14
  A brief measure of how an individual cognitively and emotionally represents their illness and its impact.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte P Malcolm, DClinPsy, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust; Faraneh Vargha-Khadem, PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irestorm E, Ora I, Linge H, Tonning Olsson I. Cognitive Fatigue and Processing Speed in Children Treated for Brain Tumours. J Int Neuropsychol Soc. 2021 Oct;27(9):865-874. doi: 10.1017/S1355617720001332. Epub 2021 Jan 14. PMID 33441219
- [Background] Patel SK, Katz ER, Richardson R, Rimmer M, Kilian S. Cognitive and problem solving training in children with cancer: a pilot project. J Pediatr Hematol Oncol. 2009 Sep;31(9):670-7. doi: 10.1097/MPH.0b013e3181b25a1d. PMID 19707159
- [Background] Butler RW, Copeland DR, Fairclough DL, Mulhern RK, Katz ER, Kazak AE, Noll RB, Patel SK, Sahler OJ. A multicenter, randomized clinical trial of a cognitive remediation program for childhood survivors of a pediatric malignancy. J Consult Clin Psychol. 2008 Jun;76(3):367-78. doi: 10.1037/0022-006X.76.3.367. PMID 18540731
- [Background] Simons DJ, Boot WR, Charness N, Gathercole SE, Chabris CF, Hambrick DZ, Stine-Morrow EA. Do "Brain-Training" Programs Work? Psychol Sci Public Interest. 2016 Oct;17(3):103-186. doi: 10.1177/1529100616661983. PMID 27697851
- [Background] Hocking MC, Paltin I, Quast LF, Barakat LP. Acceptability and Feasibility in a Pilot Randomized Clinical Trial of Computerized Working Memory Training and Parental Problem-Solving Training With Pediatric Brain Tumor Survivors. J Pediatr Psychol. 2019 Jul 1;44(6):669-678. doi: 10.1093/jpepsy/jsz015. PMID 30874803
- [Background] Treadgold B, Kennedy C, Spoudeas H, Sugden E, Walker D, Bull K. Paediatric neuro-oncology rehabilitation in the UK: carer and provider perspectives. BMJ Paediatr Open. 2019 Dec 15;3(1):e000567. doi: 10.1136/bmjpo-2019-000567. eCollection 2019. PMID 31909222
- [Background] Lassaletta A, Bouffet E, Mabbott D, Kulkarni AV. Functional and neuropsychological late outcomes in posterior fossa tumors in children. Childs Nerv Syst. 2015 Oct;31(10):1877-90. doi: 10.1007/s00381-015-2829-9. Epub 2015 Sep 9. PMID 26351237
- See also: NIHR funding awards information — https://www.dev.fundingawards.nihr.ac.uk/award/NIHR208009